CLINICAL TRIAL: NCT02477540
Title: An Open Labeled, Single-center, Phase I Study Assessing the Safety and Efficacy of Autologous Bone Marrow Derived Mesenchymal Stem Cells in Critical Limb Ischemia
Brief Title: A Safety and Efficacy Study of Autologous Bone Marrow Derived Mesenchymal Stem Cells in Critical Limb Ischemia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was stopped by sponsers internal reason.
Sponsor: Pharmicell Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cellgram-CLI
Record Dates: First submitted 2015-06-10; First posted 2015-06-22 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 2-time injection group : Cellgram-CLI (Experimental): Within 30 days after extracting bone marrow, autologous bone marrow-derived mesenchymal stem cells is directly injected into the lesion. Then the second cell is injected within 30 days after the first cell injection.
  Interventions: Drug: Cellgram-CLI

INTERVENTIONS:
Drug: Cellgram-CLI — Appearance: White cell suspension is filled in a clear plastic syringe, and fixed with an occlude on the prefilled syringe tip
  Main ingredient: Autologous bone marrow-derived mesenchymal stem cells
  Dosage: 50,000,000 cells/10ml, 2-time injection
  Storage: An airtight container, 20~25℃
  Injection Method: Intramuscular
  Other Names: Autologous bone marrow derived Mesenchymal Stem Cells

SUMMARY:
This clinical trial to study the Safety and Efficacy of Autologous Mesenchymal stem cells in critical limb ischemia.

DETAILED DESCRIPTION:
If the participant voluntarily agrees to participate in the clinical trial before registration, the investigator conducts a screening test to evaluate the participant's suitability.

A participant that satisfies all inclusion and exclusion criteria is assigned a test group(2-time injection group).

Participants conduct cell therapy within 30 days after bone marrow aspiration, and will re-inject autologous mesenchymal stem cells within 30 days after first injection.

Participants will make a total of 5 hospital visits after registration, and Safety and Efficacy will be evaluated based on a fixed procedure on every visit.

ELIGIBILITY:
Inclusion Criteria:

* Age from 20 to 80 years
* Patients with resting pain or ulceration of limb (Rutherford's class: II-4, III-5 or III-6)
* Ankle Brachial Pressure Index (ABPI) ≤ 0.6 or TCPO2 ≤ 60mmHg in the foot
* Patients who were unsuitability for percutaneous transluminal angioplasty or a bypass operation
* Patients who are not expected other treatments for at least 6 months
* Patients who can agree to participate in the clinical trial by oneself or by one's legal representative
* Patients who can conduct the clinical trial according to the protocol

Exclusion Criteria:

* Buerger's disease
* History of hematologic disease
* Patients who are at risk of embolism due to atrial fibrillation
* Primary hematologic disease, including hypercoagulable states
* Entrapment syndrome
* Patients with osteomyelitis
* Patients whose blood serum AST(Aspartate transaminase)/ALT(Alanine Transaminase) rates are more than three times the normal maximum rate, or whose creatinine rates are more than 1.5 times the normal maximum rate
* Patients with history of anaphylaxis to gentamicin
* Patients with hypersensitivity of bovine-derived ingredients
* Patients with chronic heart failure, Glomerular disease and Obstructive pulmonary disease
* Patients with Stroke or transient ischemic attack within 6 months prior to registration
* Patients tested positive for HIV(Human Immunodeficiency Virus), HCV(Hepatitis C Virus), HBV(Hepatitis B Virus) and Syphilis
* Patients with history of aorta and artery bypass operation, or angioplasty within 2 months recently
* Patients in need of a immediate amputation and have a potentially life-threatening complications of critical ischemia
* Patients with history of cell therapy
* Type I diabetes
* Uncontrolled diabetes mellitus (HgbA1C>8%)
* Uncontrolled hypertension
* Has a medical record of solid cancer, or diagnosed with solid cancer and currently receiving cancer treatment
* Positive of tumor markers test(AFP((Alpha fetoprotein), CEA(Carcinoembryonic antigen), CA15-3(Cancer antigen 15-3 for breast cancer) and PSA(Prostate-specific antigen), or have received a diagnosis of cancer based on National cancer screening program
* Pregnancy, possible candidate for pregnancy or lactating women
* Infectious disease
* Administrating of immunosuppressive agents, corticosteroid formulation and cell toxicity formulation, or requiring administration of the test period
* Patients already enrolled in another clinical trials or completed within 3 months
* Patients who cannot adapt to the protocol and follow-up observation
* Patients who has experienced drug abuse for the past 1 year
* Patients with any disease or condition which the investigator fell would interfere with trial or the safety of the subject

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Ankle Brachial Pressure Index, ABPI | 6 months after BM-MSC therapy
  Use Student's paired t-test or Wilcoxon's signed rank test to compare the difference of between the two visits(Screening and 6 month post treatment) before and after treatment.

SECONDARY OUTCOMES:
Collateral vessel formation on digital subtraction angiography (DSA) | 6 months after BM-MSC therapy
  Analyze the difference of pre and post treatment using McNemar test for homogeneity test.
Difference of Wound size | 6 months after BM-MSC therapy
  Use Student's paired t-test or Wilcoxon's signed rank test to compare the difference of pre and post treatment Healing of ulcerations (change in size of ulcers) or reduction of ulcer area in the target limb.
Improved transcutaneous oxygen pressure (TCPO2) | 6 months after BM-MSC therapy
  Use Student's paired t-test or Wilcoxon's signed rank test to compare the difference of pre and post treatment transcutaneous oxygen pressure (TCPO2).
Pain on the Visual Analogue Scale(VAS) | 6 months after BM-MSC therapy
  Use Student's paired t-test or Wilcoxon's signed rank test to compare the difference of pre and post Visual Analogue Scale(VAS).
  Visual Analogue Scale(VAS):
  Using a ruler, the score is determined by mea-suring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
  the following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm)
Reduced limb amputation | 6 months after BM-MSC therapy
  Described and define as minor amputation is below midtarsal level, major amputation is more than midtarsal level.
Temperature change on thermography | 6 months after BM-MSC therapy
  Use Student's paired t-test or Wilcoxon's signed rank test to compare the difference of pre and post thermography.
Dose about using analgesic medicine | 6 months after BM-MSC therapy
  Use Student's paired t-test or Wilcoxon's signed rank test to compare the difference between pre and post dose of the using analgesic medicine.
Change in Rutherford classification | 6 months after BM-MSC therapy
  Use Student's paired t-test or Wilcoxon's signed rank test to compare the difference of pre and post Rutherford classification.
  Rutherford classification: commonly used clinical staging system for describing peripheral arterial disease.
  Stage 0 - Asymptomatic Stage 1 - Mild claudication Stage 2 - Moderate claudication - The distance that delineates mild, moderate and severe claudication is not specified in the Rutherford classification, but is mentioned in the Fontaine classification as 200 meters.
  Stage 3 - Severe claudication Stage 4 - Rest pain Stage 5 - Ischemic ulceration not exceeding ulcer of the digits of the foot Stage 6 - Severe ischemic ulcers or frank gangrene
Frequency about using analgesic medicine | 6 months after BM-MSC therapy
  Use Student's paired t-test or Wilcoxon's signed rank test to compare the difference between pre and post frequency of the using analgesic medicine.

OTHER OUTCOMES:
For safety analysis we will observed clinical laboratory tests, physical examinations, tumor marker tests | 12 months after BM-MSC therapy
  Analyze using McNemar's test by making a table of changes that occurred in the test.
  clinical laboratory tests(Follow the unit of each institution): <Blood>
  * WBC, RBC, Hb, Hct, Platelets count, WBC Differential count, BUN, ALT, AST, Glucose, Total bilirubin, Total Cholesterol <Urine>
  * Protein, Glucose, Blood, Ketone, Billrubin, Urobillnogen
  physical examinations:
  -Allergy, Cardiovascular, Respiratory, Gastrointestinal /Liver biliary, Metabolic / endocrine, Kidney / urinary system, Reproductive, Musculoskeletal, Skin and connective, Nervous, Psyatric, Others
  tumor marker tests(Follow the unit of each institution):
  * AFP
  * CEA
  * CA15-3(female)
  * PSA(male)
occurrence and severity of adverse events | 12 months after BM-MSC therapy
  Analyze the adverse events by using seriousness, severity and relevance of IP.

CONTACTS AND LOCATIONS:
Overall Officials: WoongChol Kang, MD, Ph.D, Principal Investigator — Gachon University Gil Medical Center